CLINICAL TRIAL: NCT05344638
Title: A Multicenter, Randomized, Double-Blind, Parallel, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of AGS Compared to AGU for Acute Bronchitis
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of "AG1904" in Acute Bronchitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AG1904
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Acute Bronchitis
MeSH Terms: conditions — Bronchitis | interventions — Aspartylglucosylaminase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AGS (Experimental) (Experimental): AGS + Placebo of AGU
  Interventions: Drug: AGS (Experimental)
- AGU (Active Comparator) (Active Comparator): Placebo of AGS + AGU
  Interventions: Drug: AGU (Active Comparator)

INTERVENTIONS:
Drug: AGS (Experimental) — tid
  Arms: AGS (Experimental)
Drug: AGU (Active Comparator) — tid
  Arms: AGU (Active Comparator)

SUMMARY:
A Multicenter, Randomized, Double-Blind, Parallel, Active-controlled, Phase III Clinical Trial to Evaluate the Efficacy and Safety of AGS Compared to AGU for Acute Bronchitis

ELIGIBILITY:
Inclusion Criteria:

* Both gender, 19 years ≤ age ≤ 75 years
* BSS(Bronchitis Severity Score) ≥ 5point at Visit 2 (Randomized Visit)
* Patients without fever based on Visit 2(Randomized Visit)
* Those who can comply with the requirements of clinical trials
* Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

* Patients with respiratory and systemic infections requiring systemic antibiotic therapy
* Patients with bleeding tendency or coagulation disorder
* Patients who investigators determines to severe respiratory disease that would interfere with study assessment
* Those who have participated in other clinical trials within 4 weeks before participating in clinical trials
* In case the investigator judges that it is not suitable for the subject of this clinical trial for other reasons

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Bronchitis Severity Total Score(BSS) change of Visit 3 compared to Visit 2 | Visit 1 (-3 day), Visit 2 (0 day), Visit 3 (7 day)
  The BSS comprises the following five symptoms typical for Acute Bronchitis: cough, sputum, rales/rhonchi on auscultation, chest pain during coughing, and dyspnea. These symptoms are each assessed according to a 5-point scale: 0 = absent, 1 = mild, 2 = moderate, 3 = severe and 4 = very severe

SECONDARY OUTCOMES:
Individual symptom score of Bronchitis Severity Score(BSS) of Visit 3 compared to Visit 2 | 7days
Treatment response rate at Visit 3 | 7days
Integrative Medicine Outcome Scale (IMOS) | 7days
Integrative Medicine Patient Satisfaction Scale (IMPSS) | 7days

CONTACTS AND LOCATIONS:
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea